CLINICAL TRIAL: NCT03528772
Title: Topical 5% Minoxidil Versus 0.2%Topical Glyceryl Trinitrate in Treatment of Chronic Anal Fissure: a Randomized Controlled Trial
Brief Title: Topical Minoxidil Versus Topical Glyceryl Trinitrate in Treatment of Chronic Anal Fissure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Lecturer of general surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: mansoura50
Record Dates: First submitted 2018-05-06; First posted 2018-05-18 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Anal Fissure
Keywords: anal fissure, minoxidil, glycreyl trinitrate
MeSH Terms: conditions — Fissure in Ano | interventions — Minoxidil; Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minoxidil (Active Comparator): Patients in this arm will receive topical treatment with Minoxidil forte 5% gel three times per days for 4 weeks
  Interventions: Drug: Minoxidil
- Glyceryl trinitrate (Active Comparator): Patients in this arm will receive topical treatment with glyceryl trinitrate 0.2% cream three times per days for 4 weeks
  Interventions: Drug: Glyceryl trinitrate

INTERVENTIONS:
Drug: Minoxidil — application of minoxidil forte 5% gel three time per day on the anus for four weeks
  Other Names: Topical Minoxidil treatment
  Arms: Minoxidil
Drug: Glyceryl trinitrate — application of glyceryl trinitrate 0.2% cream three time per day on the anus for four weeks
  Other Names: Topical GTN treatment
  Arms: Glyceryl trinitrate

SUMMARY:
This randomized trial aims to compare two topical treatments in the treatment of chronic anal fissure: minoxidil gel and glycreyl trintrate cream. The endpoint of the study is the duration of healing of anal fissure whereas secondary endpoints include adverse effects of each treatment and recurrence of anal fissure

DETAILED DESCRIPTION:
All participants who fulfill the inclusion criteria and give consent for participation in the trial and will be included and randomly assigned to either group I (5% Minoxidil gel) or group II (0.2% GTN cream) with a 1:1 allocation. Randomization will be carried out using online software (Research Randomizer Version 4.0 at https://www.randomizer.org).

Patients will receive the topical agent in unlabeled red or blue containers. The code of each color will be known to a pharmacist who will not take any part in patients' care, follow-up, data collection/analysis or accessing outcomes of the study. The investigators will be blinded to the nature of content of each container and the outcome assessor will not be aware of the study nature.

Interventions Eligible patients will be randomized into two equal groups: groups I will receive topical 5% Minoxidil gel (Minoxidil Forte 5% topical gel 60 gm; Pharmacare Egypt Co., Cairo, Egypt) and group II will receive topical 0.2% GTN cream (Nitoglycerine-Glycerile Tinitrade 0.2%, 30 gm; E.S.A.G Pharma Co., Cairo, Egypt). Both agents used in the study will be relabeled by a pharmacist who will not take any part in the study in terms of patients' care, follow-up, data collection/analysis or accessing outcomes. Both topical agents will be placed in identical containers of 60 gm and labeled with blue or red colors. The color code will remain undefined till the end of trial, data analysis, and interpretation of results except for the same pharmacist. The containers will be distributed to the patients by the outpatient's department nurse in the hospital.

Patients will be advised to apply approximately 2 cm of the gel/cream (equal to 3 gm) on the perianal area three times per day for 4 weeks. The first dose of drugs will be given at home on the same day of the first visit. During the first visit, patients will be taught to self-administer the topical gel/cream. The patients will be instructed to take laxatives to avoid constipation and to avoid using other topical preparations during the study period.

Follow-up Patients will be followed in the general and colorectal surgery outpatient clinics for a period of three months. Patients will be advised to visit the outpatient clinic every week for one month, then biweekly in the 2nd and 3rd months after starting treatment. In case of intolerable adverse events patients will be advised to visit the outpatient clinic at any other time point during the trial. At each visit the anal fissure will be inspected and the extent of healing will be assessed by a surgical resident who is unaware of the nature of the study. Patients will be asked about the improvement in their symptoms, particularly anal pain and bleeding. Pain will be measured at each visit by the Visual Analog Scale (VAS) ranging from no pain "0" to worst possible pain "10". Blood pressures will be measured and any decrease of > 15 mmHg from the basal pressure measured at the first visit will be considered significant. Adverse effects induced by the topical agents as itching, headache, palpitation, dizziness, excess perianal hair growth, and hypersensitivity reaction will be recorded. Itching will be assessed by 5-D pruritus scale. The continence state will be assessed using Wexner continence score.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders presenting with chronic anal fissure of more than 6 weeks in duration
* Ageing between 18 and 65 years old.

Exclusion Criteria:

* Pregnant patients.
* Patients with recurrent anal fissure after previous sphincterotomy.
* Patients with coexisting anorectal diseases or inflammatory bowel diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Healing duration | two months
  the duration of time needed for complete healing defined as reepithelialization of the anoderm at the site of anal fissure

SECONDARY OUTCOMES:
Anal pain | three months
  degree of relief of anal pain as measured by visual analogue scale (VAS) from 0 to 10 where 0 indicates no pain and 10 indicates the worst severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Emile, M.D., Principal Investigator — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Emile SH, Abdel-Razik MA, Elshobaky A, Elbaz SA, Khafagy W, Shalaby M. Topical 5% minoxidil versus topical 0.2% glyceryl trinitrate in treatment of chronic anal fissure: A randomized clinical trial. Int J Surg. 2020 Mar;75:152-158. doi: 10.1016/j.ijsu.2020.01.143. Epub 2020 Feb 4. PMID 32028023